CLINICAL TRIAL: NCT05944705
Title: Commercially Available Cannabis (Hemp) Products for Immune Support: A Prospective Observational Study to Evaluate Safety and Effects
Brief Title: Commercially Available Cannabis Products for Immune Support
Status: Recruiting | Type: Observational
Sponsor: Center For Interventional Pain and Spine (Other)
Collaborators: Agronomed LLC (Unknown)
Responsible Party: Sponsor
Other Study IDs: CannabisforImmuneSupport
Record Dates: First submitted 2023-02-20; First posted 2023-07-13 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Influenza; COVID-19; Common Cold
MeSH Terms: conditions — Influenza, Human; COVID-19; Common Cold

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Symptomatic individuals using hemp or cannabis products for immune support: Individuals with symptomatic illness that utilize a proprietary hemp or cannabis product to aid in their recovery
  Interventions: Dietary Supplement: Immune Support Supplement
- Symptomatic individuals not currently using hemp or cannabis products for immune support: Individuals without symptomatic illness that do not utilize the proprietary hemp or cannabis product to aid in their recovery

INTERVENTIONS:
Dietary Supplement: Immune Support Supplement — Cannabinoid and co-active emulsion
  Groups: Symptomatic individuals using hemp or cannabis products for immune support

SUMMARY:
This study will be a prospective observation of the use of commercially available hemp and cannabis products marketed for immune support.

DETAILED DESCRIPTION:
In the era of COVID-19, there has been much speculation about the risks and benefits of cannabis use for immune support. It is well known that the endocannabinoid system plays a role in the regulation of the immune response and its role in inflammation reduction may be useful in terms of a potential adjunctive therapy for acute infection. Cannabis products vary widely in their composition and may have a varying effect based on the strain and the associated terpenes. Here, we aim to track cannabis and hemp usage during an acute infection to understand it's safety and effects in a symptomatic population.

Given the fast and widespread acceptance and use of cannabis products in the US market, commercial use has outpaced randomized controlled trials (RCTs). Thus, carefully designed observational studies are important to understand how these products are affecting consumers. Prospective observational designs allow for real-world examinations of commercialized products with similar effect sizes to RCTs. Although observational designs have some drawbacks, a review covering 1,583 meta-analyses across 228 medical conditions compared the effect sizes from RCTs with those from observational studies for the same medical conditions and found no differences between the two. (1) These data provide evidence that a carefully designed observational study can help us better understand the effects of commonly used products such as cannabis edibles. The aim of this observational study is to evaluate the safety and associated effects of commercially available cannabis products in the US in symptomatic individuals seeking them for immune support.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able to read and write in English
3. Active participants in the Pennsylvania medical marijuana program (for cannabis product users)
4. Currently experiencing one or more of the following symptoms due to an acute illness:

   1. Fever or chills
   2. Cough
   3. Fatigue
   4. Muscle or body aches
   5. Headache
   6. Sore throat
   7. Congestion or runny nose
   8. Nausea or Vomiting
   9. Diarrhea
5. Agrees to consume their chosen hemp or cannabis product (for the cannabis arm) and to not use a different hemp or cannabis product through the duration of the study
6. Agrees to continue to abstain from using hemp or cannabis (for the non-cannabis/hemp using arm)
7. Must have smart phone or email and access to the internet
8. Be able to comply with study requirements including baseline, completion of electronic questionnaires, and study timeline parameters.

Exclusion Criteria:

1. Women who are pregnant, breastfeeding, or planning to become pregnant.
2. Known allergy to any compounds in hemp or cannabis.
3. Endorses suicidal intent
4. Immunocompromised individuals
5. Unwilling or unable to comply with study procedures
6. Terminal Illness with life expectancy less than 1 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals who are suffering an acute illness
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2024-11-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Eventss | To Study Completion, approximately 30 days
  Evaluate the safety of commercially available hemp and cannabis products marketed for immune support through assessment of AEs and SAEs. AEs and SAEs will also be collected for the non-user group

SECONDARY OUTCOMES:
Symptom Improvement | 3 days
  Quantify subject-reported changes in symptoms during the course of their illness at baseline, 3-, 5-, 10- 15- and 30-days via electronic survey collection.
Symptom Improvement | 5 days
  Quantify subject-reported changes in symptoms during the course of their illness at baseline, 3-, 5-, 10- 15- and 30-days via electronic survey collection.
Symptom Improvement | 10 days
  Quantify subject-reported changes in symptoms during the course of their illness at baseline, 3-, 5-, 10- 15- and 30-days via electronic survey collection.
Symptom Improvement | 15 days
  Quantify subject-reported changes in symptoms during the course of their illness at baseline, 3-, 5-, 10- 15- and 30-days via electronic survey collection.
Symptom Improvement | 30 days
  Quantify subject-reported changes in symptoms during the course of their illness at baseline, 3-, 5-, 10- 15- and 30-days via electronic survey collection.
Profile of Mood States (POMS) | 3 days
  The Profile of Mood States is a subject-reported questionnaire that measures the six different dimensions of mood swings. These dimensions include tension or anxiety, anger or hostility, vigor or activity, fatigue or inertia, depression or dejection, confusion or bewilderment. This scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). Higher scores on the POMS subscales reflect a greater agreement with the mood state during the past week.
Profile of Mood States (POMS) | 5 days
  The Profile of Mood States is a subject-reported questionnaire that measures the six different dimensions of mood swings. These dimensions include tension or anxiety, anger or hostility, vigor or activity, fatigue or inertia, depression or dejection, confusion or bewilderment. This scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). Higher scores on the POMS subscales reflect a greater agreement with the mood state during the past week.
Profile of Mood States (POMS) | 10 days
  The Profile of Mood States is a subject-reported questionnaire that measures the six different dimensions of mood swings. These dimensions include tension or anxiety, anger or hostility, vigor or activity, fatigue or inertia, depression or dejection, confusion or bewilderment. This scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). Higher scores on the POMS subscales reflect a greater agreement with the mood state during the past week.
Profile of Mood States (POMS) | 15 days
  The Profile of Mood States is a subject-reported questionnaire that measures the six different dimensions of mood swings. These dimensions include tension or anxiety, anger or hostility, vigor or activity, fatigue or inertia, depression or dejection, confusion or bewilderment. This scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). Higher scores on the POMS subscales reflect a greater agreement with the mood state during the past week.
Profile of Mood States (POMS) | 30 days
  The Profile of Mood States is a subject-reported questionnaire that measures the six different dimensions of mood swings. These dimensions include tension or anxiety, anger or hostility, vigor or activity, fatigue or inertia, depression or dejection, confusion or bewilderment. This scale contains 65 self-report items using the 5-point Likert Scale. Participants can choose from 0 (not at all) to 4 (extremely). Higher scores on the POMS subscales reflect a greater agreement with the mood state during the past week.
Quality of Life and Sleep via Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 3 days
  The Subject-Reported Outcomes Measurement Information System is a questionnaire that assesses pain intensity in addition to several correlating domains of health. The domains of health assessed include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Quality of Life and Sleep via Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 5 days
  The Subject-Reported Outcomes Measurement Information System is a questionnaire that assesses pain intensity in addition to several correlating domains of health. The domains of health assessed include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Quality of Life and Sleep via Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 10 days
  The Subject-Reported Outcomes Measurement Information System is a questionnaire that assesses pain intensity in addition to several correlating domains of health. The domains of health assessed include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Quality of Life and Sleep via Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 15 days
  The Subject-Reported Outcomes Measurement Information System is a questionnaire that assesses pain intensity in addition to several correlating domains of health. The domains of health assessed include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Quality of Life and Sleep via Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 30 days
  The Subject-Reported Outcomes Measurement Information System is a questionnaire that assesses pain intensity in addition to several correlating domains of health. The domains of health assessed include physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance. The patients' answers to the PROMIS-29 are scored from 1-5 (with the exception of the NRS). The sum of the PROMIS results in the raw score, which lies between 4 and 20. There is no total score, but each axis forms its own score.
Time back to work/normal activities | 3 days
  Average time back to work/normal activities will be measured by collecting the day at which the individual became ill and missed work/normal activities and collecting the day at which work/normal activities will be resumed.
Time back to work/normal activities | 5 days
  Average time back to work/normal activities will be measured by collecting the day at which the individual became ill and missed work/normal activities and collecting the day at which work/normal activities will be resumed.
Time back to work/normal activities | 10 days
  Average time back to work/normal activities will be measured by collecting the day at which the individual became ill and missed work/normal activities and collecting the day at which work/normal activities will be resumed.
Time back to work/normal activities | 15 days
  Average time back to work/normal activities will be measured by collecting the day at which the individual became ill and missed work/normal activities and collecting the day at which work/normal activities will be resumed.
Time back to work/normal activities | 30 days
  Average time back to work/normal activities will be measured by collecting the day at which the individual became ill and missed work/normal activities and collecting the day at which work/normal activities will be resumed.
Concomitant medications and supplements | To Study Completion, approximately 30 days
  All medications taken over the course of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Philip Kim, MD, Principal Investigator — Center For Interventional Pain and Spine
Locations (1):
- Center for Interventional Pain and Spine, Bryn Mawr, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No